CLINICAL TRIAL: NCT04380974
Title: A Random, Open-label Multicenter, Phase IV Study Assessing the Efficacy and Safety of Two Regimens of Anti-VEGF Therapy in Chinese Patients With Polypoidal Choroidal Vasculopathy
Brief Title: Efficacy and Safety of Two Regimens of Anti-VEGF Therapy in Chinese Patients With Polypoidal Choroidal Vasculopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaodong Sun (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaodong Sun, Professor and Executive Vicechair of Department of Ophthalmology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCV20200506
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal Choroidal Vasculopathy; Optical coherence tomography angiography; Optical coherence tomography
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCTA plus OCT guided 3+PRN regimen (Experimental): Monthly intravitreal injections of anti-VEGF drug in the core treatment period and PRN intravitreal injections of the same dose guided by BCVA stabilization, OCTA and OCT in the extension treatment period.
  Interventions: Procedure: OCTA plus OCT guided 3+PRN regimen; Drug: Anti-VEGF drug
- OCT guided 3+PRN regimen (Active Comparator): Monthly intravitreal injections of anti-VEGF drug in the core treatment period and PRN intravitreal injections of the same dose guided by BCVA stabilization and OCT in the extension treatment period.
  Interventions: Procedure: OCT guided 3+PRN regimen; Drug: Anti-VEGF drug

INTERVENTIONS:
Procedure: OCTA plus OCT guided 3+PRN regimen — For the OCTA plus OCT guided 3+PRN regimen, we recorded patients' data after retreatment by 3 monthly intravitreal injections of anti-VEGF drug. Subsequent reinjections were given as needed according to the changes in patients' visual acuity, activity of PCV lesions shown by OCTA and/or the exudation shown by OCT. Four weeks after the third and last injection, all patients in this group underwent an examination, including ETDRS visual acuity, fundus photography, OCTA and OCT.
  In case of BVN increased or polypoidal lesion progressed on OCTA scans, persistent subfoveal or perifoveal fluid, macular intraretinal edema on OCT scans, or visual loss of >5 letters, or the occurrence of a new hemorrhage, patients were retreated. The persistence of hemorrhage without evidence of fluid was not considered a criterion for retreatment. In the absence of retreatment criteria, no further injections were given and another examination was proposed usually 4 weeks later.
  Arms: OCTA plus OCT guided 3+PRN regimen
Procedure: OCT guided 3+PRN regimen — For the OCT guided 3+PRN group, we recorded patients'data after retreatment by 3 monthly intravitreal injections of Anti-VEGF drugs. Subsequent reinjections were given as needed according to the changes in patients'visual acuity and/or the exudation shown by OCT. Four weeks after the third and last injection, all patients in this group underwent an examination, including ETDRS visual acuity, fundus photography, and OCT.
  In case of persistent subfoveal or perifoveal fluid, macular intraretinal edema, visual loss of >5 letters, or the occurrence of a new hemorrhage, patients were retreated. The persistence of hemorrhage without evidence of fluid was not considered a criterion for retreatment. In the absence of retreatment criteria, no further injections were given and another examination was proposed usually 4 weeks later.
  Arms: OCT guided 3+PRN regimen
Drug: Anti-VEGF drug — Conbercept or other anti-VEGF drugs

SUMMARY:
The study will evaluate the efficacy and safety of two different regimens of anti-VEGF Therapy (OCTA plus OCT guided 3+PRN vs. OCT guided 3+PRN) in Chinese patients with PCV. This study is to provide long-term safety data in the treatment of Chinese patients with PCV.

ELIGIBILITY:
Inclusion Criteria:

* Written informed-consent before any evaluation
* Visual impairment due to PCV, including type 1 PCV and type 2 PCV.
* 50 years old and older
* Chinese
* For study eye: BCVA between 20/30 and 20/320 on electronic visual acuity texting at the time point of both screening and baseline.

Exclusion Criteria:

* Have Stroke and myocardial infarction within 3 months before screening
* Any active periocular and ocular infection and inflammation (including blepharitis, conjunctivitis, keratitis, scleritis, uveitis, intraocular inflammation) while screening and baseline.
* Uncontrolled glaucoma (under treatment [IOP] ≥ 30 mm Hg or depend on researchers) while screening and baseline
* Neovascularization of iris and neovascular glaucoma while screening and baseline
* Any causes led to choroidal neovascularization except PCV (including ICNV, central serous chorioretinopathy, ocular histoplazmoza and pathologic myopia) while screening and baseline
* With structure injury (including vitreous macular traction,epiretinal membrane involving in central fovea,subretinal fibroplasia,laser scar and central fovea atrophy) within 0.5 optic disc diameter to the central of macula while screening and baseline, which may harm the improvement of vision by treatment according to researchers
* Any systemic anti-VEGF medication(as Avastin) use within 3 months before screening
* Any medication systemic use toxic to lens, retina and optic nerve, including iron amine, chloroquine/chloroquine (Plaquenil ®), tamoxifen, phenothiazine and ethambutol
* For study eye: Used to accept following treatments for PCV within 3 months or accept following treatments more than three times before baseline:

  1. Anti-angiogenesis drugs (pegaptanib, ranibizumab, bevacizumab),VEGF-Trap;
  2. Anecortave acetate corticosteroids;
  3. Protein kinase C inhibitors, squalamine, siRNA;
  4. PDT, Visudyne® treatment, external beam radiotherapy, local laser photocoagulation, vitrectomy, submacular surgery and transpupillary thermotherapy
* Any intraocular surgery (including YAG laser) within 3 months before baseline or predicated within 6 months after baseline
* Intraocular or periocular treatment of corticosteroids within 3 months before baseline
* For follow eye: Any anti-angiogenesis treatment (including anti-VEGF, like Lucentis, Avastin and KH902 ) within 3 months before baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
PCV lesion recurrence | 24 months
  PCV lesion recurrence is defined as the reappearance of new exudative biomakers (such as IRF, SRF, PED) or new hemorrhage detected on OCT or fundus examination in subsequent visits from the last visit showing clinical stability. PCV lesion recurrence rate will be compared at 24months between the two groups to assess the efficacy of OCTA plus OCT guided 3+PRN regimen.

SECONDARY OUTCOMES:
Mean Snellen BCVA at every visit or treatment | 24 months
  Compare of mean Snellen Best-Corrected-visual-acuity at every visit or treatment between the two groups to assess the efficacy of OCTA plus OCT guided 3+PRN regimen.
Number of participants with treatment-related adverse events | 24 months
  Compare of Number of participants with treatment-related adverse events between the two groups to assess the safety of OCTA plus OCT guided 3+PRN regimen
Mean number of injections after the initial three loading dose monthly injections | 21 months
  Compare of mean number of injections after the initial three loading dose monthly injections between the two groups to assess the efficacy of OCTA plus OCT guided 3+PRN regimen.
Mean central macular thickness at every visit or treatment by OCT | 24 months
  Compare of mean central macular thickness by OCT at every visit or treatment between the two groups to assess the efficacy of OCTA plus OCT guided 3+PRN regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yannuzzi LA, Sorenson J, Spaide RF, Lipson B. Idiopathic polypoidal choroidal vasculopathy (IPCV). 1990. Retina. 2012 Feb;32 Suppl 1:1-8. PMID 22451948
- [Background] Cheung CMG, Lai TYY, Ruamviboonsuk P, Chen SJ, Chen Y, Freund KB, Gomi F, Koh AH, Lee WK, Wong TY. Polypoidal Choroidal Vasculopathy: Definition, Pathogenesis, Diagnosis, and Management. Ophthalmology. 2018 May;125(5):708-724. doi: 10.1016/j.ophtha.2017.11.019. Epub 2018 Jan 10. PMID 29331556
- [Background] Wong CW, Yanagi Y, Lee WK, Ogura Y, Yeo I, Wong TY, Cheung CMG. Age-related macular degeneration and polypoidal choroidal vasculopathy in Asians. Prog Retin Eye Res. 2016 Jul;53:107-139. doi: 10.1016/j.preteyeres.2016.04.002. Epub 2016 Apr 14. PMID 27094371
- [Background] Marcus DM, Singh H, Lott MN, Singh J, Marcus MD. Intravitreal ranibizumab for polypoidal choroidal vasculopathy in non-Asian patients. Retina. 2013 Jan;33(1):35-47. doi: 10.1097/IAE.0b013e3182618be0. PMID 22990319
- [Background] Cho HJ, Koh KM, Kim HS, Lee TG, Kim CG, Kim JW. Anti-vascular endothelial growth factor monotherapy in the treatment of submacular hemorrhage secondary to polypoidal choroidal vasculopathy. Am J Ophthalmol. 2013 Sep;156(3):524-531.e1. doi: 10.1016/j.ajo.2013.04.029. Epub 2013 Jun 13. PMID 23769197
- [Background] Cheung CM, Li X, Mathur R, Lee SY, Chan CM, Yeo I, Loh BK, Williams R, Wong EY, Wong D, Wong TY. A prospective study of treatment patterns and 1-year outcome of Asian age-related macular degeneration and polypoidal choroidal vasculopathy. PLoS One. 2014 Jun 30;9(6):e101057. doi: 10.1371/journal.pone.0101057. eCollection 2014. PMID 24978485
- [Background] Hikichi T, Higuchi M, Matsushita T, Kosaka S, Matsushita R, Takami K, Ohtsuka H, Ariga H. One-year results of three monthly ranibizumab injections and as-needed reinjections for polypoidal choroidal vasculopathy in Japanese patients. Am J Ophthalmol. 2012 Jul;154(1):117-124.e1. doi: 10.1016/j.ajo.2011.12.019. Epub 2012 Apr 1. PMID 22465366
- [Background] Hikichi T, Higuchi M, Matsushita T, Kosaka S, Matsushita R, Takami K, Ohtsuka H, Kitamei H, Shioya S. Results of 2 years of treatment with as-needed ranibizumab reinjection for polypoidal choroidal vasculopathy. Br J Ophthalmol. 2013 May;97(5):617-21. doi: 10.1136/bjophthalmol-2012-302652. Epub 2013 Feb 21. PMID 23428984
- [Background] Kang HM, Koh HJ. Long-term visual outcome and prognostic factors after intravitreal ranibizumab injections for polypoidal choroidal vasculopathy. Am J Ophthalmol. 2013 Oct;156(4):652-60. doi: 10.1016/j.ajo.2013.05.038. Epub 2013 Jul 24. PMID 23891333
- [Background] Inoue M, Balaratnasingam C, Freund KB. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY OF POLYPOIDAL CHOROIDAL VASCULOPATHY AND POLYPOIDAL CHOROIDAL NEOVASCULARIZATION. Retina. 2015 Nov;35(11):2265-74. doi: 10.1097/IAE.0000000000000777. PMID 26405770
- [Background] Wang M, Zhou Y, Gao SS, Liu W, Huang Y, Huang D, Jia Y. Evaluating Polypoidal Choroidal Vasculopathy With Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT526-32. doi: 10.1167/iovs.15-18955. PMID 27472276
- [Background] Chan SY, Wang Q, Wang YX, Shi XH, Jonas JB, Wei WB. POLYPOIDAL CHOROIDAL VASCULOPATHY UPON OPTICAL COHERENCE TOMOGRAPHIC ANGIOGRAPHY. Retina. 2018 Jun;38(6):1187-1194. doi: 10.1097/IAE.0000000000001702. PMID 28613216
- [Background] Bo Q, Yan Q, Shen M, Song M, Sun M, Yu Y, Rosenfeld PJ, Wang F, Sun X. Appearance of Polypoidal Lesions in Patients With Polypoidal Choroidal Vasculopathy Using Swept-Source Optical Coherence Tomographic Angiography. JAMA Ophthalmol. 2019 Jun 1;137(6):642-650. doi: 10.1001/jamaophthalmol.2019.0449. PMID 30998817